CLINICAL TRIAL: NCT03896529
Title: Neurobiological Mechanisms of Aging and Stress on Prospective Navigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H18233; R21AG063131 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Aging; Anxiety; Memory Impairment
Keywords: Aging; Spatial Memory; Stress; fMRI
MeSH Terms: conditions — Anxiety Disorders; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Behavioral (Psychological stress manipulation). Between-subjects design. Participants will be assigned to either a stress-manipulated or control (no stress induced) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-stress control group (No Intervention): Participants in this group will perform the psychology tasks (virtual navigation) without any manipulation of psychological stress
- Stress group (Experimental): Participants in this group will perform the psychology tasks (virtual navigation) under manipulated psychological stress (anticipatory threat of shock)
  Interventions: Behavioral: Anticipatory psychological stress

INTERVENTIONS:
Behavioral: Anticipatory psychological stress — Unpredictable delivery of low-level electrical stimulation to left ankle periodically throughout psychology tasks (virtual navigation). Established procedure for inducing anticipatory stress.
  Arms: Stress group

SUMMARY:
Two hallmarks of both healthy aging and age-related disease are 1) memory and navigational deficits, particularly in orienting towards goal locations and planning how to navigate to them, and 2) increased susceptibility to stress and altered regulation of the stress response. However, there are marked individual differences in these age-related changes. The investigators' proposal will help characterize factors that contribute to this variability.

Participants will be pseudorandomly assigned to stress-manipulated or control groups. The investigators will give both groups a novel immersive navigation task, validated by the PI in healthy young adults. This paradigm gives participants the opportunity to either (a) flexibly draw on spatial memory in order to plan efficient routes to goal locations, or (b) fall back on inefficient, but cognitively less-demanding, stimulus-response associations (i.e., habits). Using neuroimaging and behavioral measures, the investigators' protocol will test whether experimentally-induced stress leads individuals to bring fewer details about future locations to mind when route planning, and whether such restricted prospective thought ultimately biases participants towards relatively inflexible, habitual actions.

DETAILED DESCRIPTION:
Two hallmarks of both healthy aging and age-related disease are 1) memory and navigational deficits, particularly in orienting towards goal locations and planning how to navigate to them, and 2) increased susceptibility to stress and altered regulation of the stress response. However, there are marked individual differences in these age-related changes. The investigators' proposal will help characterize factors that contribute to this variability.

The investigators propose a study that utilizes cutting-edge imaging and virtual reality techniques to characterize the neural mechanisms of prospective (future goal-directed) navigational planning in aging. The investigators will use multi-voxel pattern analyses (MVPA) to obtain neural indices of memory-guided navigational planning. The investigators will then examine the mechanisms through which stress limits the ability of individuals to flexibly navigate to future goals. A critical aim will be to evaluate the neural bases for individual differences in navigational planning and the stress response, providing novel insight into convergent neurocognitive traits that underlie different degrees of age-related cognitive decline. The investigators predict that impaired prospective planning is associated with individual differences in (a) susceptibility to exogenous, experimentally-induced stress, and (b) stress-disrupted functioning of memory and attention and cognitive control networks necessary for mental simulation.

The investigators' proposal combines a novel immersive navigation paradigm, validated by the PI in healthy young adults, and an established between-subjects exogenous manipulation of psychological stress (see Research Strategy). This paradigm gives participants the opportunity to either (a) flexibly draw on spatial memory in order to plan efficient routes to goal locations, or (b) fall back on inefficient, but cognitively less-demanding, stimulus-response associations (i.e., habits). Participants will be pseudorandomly assigned to stress-manipulated or control groups, with an initial prospective random assignment of subject IDs being adjusted as recruitment progresses in order to enforce approximately equivalent age distributions in the two groups (and thus limit confounds in subsequent group comparisons). Salivary cortisol (stress hormone) assays (de-identified) will help validate the stress difference between groups. Leveraging MVPA, and trait questionnaires, the investigators' study will test whether experimentally-induced stress leads individuals to bring fewer details about future locations to mind when route planning, and whether such restricted prospective thought ultimately biases participants towards relatively inflexible, habitual actions.

Aging is associated with differences in the degree to which people rely on "map-like" spatial memory vs. procedural motor responses to traverse environments. Thus the investigators' investigation of the effects of stress on habitual vs. prospective spatial memory-guided navigation is embedded within the context of age-related differences in spatial memory processing in the investigators' target population. The investigators will further employ an endogenous navigational strategy identification task, enabling us to 1) establish a link between endogenous navigation strategy preferences and performance on the investigators' prospective navigation task, and 2) study how endogenous navigational strategy preferences interact with induced stress to affect the investigators' neural and behavioral outcome measures indexing efficient, prospective spatial cognition.

ELIGIBILITY:
Inclusion Criteria:

* adults 65-80
* U.S. citizens or permanent residents
* who speak fluent English
* willing to come to Georgia Tech to participate in group testing sessions.

Exclusion Criteria:

* Individuals will be carefully screened using IRB-approved procedures for safety contraindications to MRI and electrical shock stimulation
* (e.g., metal or electrical implants, heart arrhythmia, or medication affecting the cardiovascular system [e.g. beta-blockers]).

The purpose of this study is to investigate mechanisms of normally functioning memory, and memory-related changes in healthy aging. Thus, any confounding factors that may influence cognition, other than age, will be exclusionary. Potential participants that endorse any of the following conditions will be excluded from the study:

* Epilepsy
* Dementia
* Parkinson's disease
* history of stroke or seizure
* psychiatric disorders
* untreated depression or emotional conditions
* Attention Deficit Disorder
* Multiple Sclerosis
* uncontrolled hyper- or hypo-tension
* untreated Diabetes
* Sickle Cell Anemia
* regularly use illegal or psychoactive drugs (e.g., cocaine, alcohol abuse, etc).
* Additionally, individuals scoring < 3 on WAIS-R forward span, < 2 on WAIS-R backward span, and failing to name more than 2 vegetable names will be excluded from the study. These exclusions will insure that persons with mild cognitive impairment or typical indications of clinical dementia will be not participate in the research.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral probability of taking a shortcut between control and treatment groups | Approximately 1.5 years
  Probability of taking a virtual navigation shortcut on an fMRI task trial, compared between stress and control groups. Measurement tool: objective categorical measure (no scale) reflecting proportion of trials in which participants traverse the shortcut road or, alternatively, the familiar (longer) road in a virtual environment.
fMRI activation level between control and treatment groups | Approximately 1.5 years
  Network activation levels (across frontoparietal, hippocampal, and striatal memory network) during fMRI task trials, compared between stress and control groups. Measurement tool: fMRI activity level. Scale: continuous activity level estimates from fMRI.
Neural memory representation reactivation between control and treatment groups | Approximately 1.5 years
  Memory reactivation levels in neural activity patterns during fMRI task, compared between stress and control groups. Measurement tool: Machine learning algorithm trained to decode fMRI patterns across voxels. Scale: algorithm success at classifying fMRI patterns according to the correct location memory for a given fMRI task trial

SECONDARY OUTCOMES:
Relationship between fMRI activity level and behavioral probability of taking a shortcut. | Approximately 1.5 years
  A linear regression will relate continuous network activity levels (Outcome measure 2) across participants with proportion of virtual navigation shortcuts (shortcut vs familiar route; Outcome measure 1). Measurement tool: fMRI and objective categorical measure of route choice behavior during fMRI task.
2. Salivary cortisol (stress hormone) response difference between stress and control participant groups. | Approximately 1.5 years
  A two-sample t-test will compare stress hormone levels (cortisol from saliva sample) between the stress and control groups. Measurement tool: cotton swab (salivette) assay of de-identified hormone levels in saliva during fMRI task.

CONTACTS AND LOCATIONS:
Overall Officials: Thackery I Brown, Ph.D., Principal Investigator — Georgia Institute of Technology
Locations (1):
- Center for Advance Brain Imaging, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No